CLINICAL TRIAL: NCT00895453
Title: Monthly Itraconazole Versus Classic Homeopathy for the Treatment of Recurrent Vulvovaginal Candidiasis: a Randomised Trial
Brief Title: Monthly Itraconazole Versus Classic Homeopathy for Treatment of Recurrent Vulvovaginal Candidiasis (RVVC)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Armin Witt, Vienna Medical School
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 134/2000
Record Dates: First submitted 2009-01-16; First posted 2009-05-08 (Estimated); Results first posted 2009-05-08 (Estimated); Last update posted 2016-11-11 (Estimated); Status verified 2009-05

CONDITIONS: Vulvovaginal Candidiasis
Keywords: recurrent vulvovaginal candidiasis; itraconazole; classic homeopathy
MeSH Terms: conditions — Candidiasis, Vulvovaginal | interventions — Itraconazole; 6-phospho-beta-galactosidase; Iron, Dietary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- itraconazole (Active Comparator): 6-months maintenance regimen with monthly single-day itraconazole 200mg twice daily (bid).
  Interventions: Drug: itraconazole
- itraconazole + lactobacilli agent (Active Comparator): 6-months maintenance regimen with monthly single-day itraconazole 200mg twice daily (bid). Additionally, Lactobacillus vaginal tablets monthly given through 6 days.
  Interventions: Drug: itraconazole; Drug: lactobacillus gasseri
- classic homeopathy (CH) (Active Comparator): CH treatment was provided by a licensed CH practitioner. Specifically, a personal history was taken and an individualised treatment scheme was prescribed. The most often used homeopathic remedies were carcinosin M, nux vomica, pulsatilla M, ferrum metallicum, and sepia M. Potencies of homeopathic remedies ranged from C 30 to C 1000.
  Interventions: Drug: classic homeopathy (carcinosin M, nux vomica, pulsatilla M, ferrum metallicum, sepia M, etc. as prescribed)

INTERVENTIONS:
Drug: itraconazole — 6-months maintenance regimen with monthly single-day itraconazole 200mg twice daily (bid)
  Arms: itraconazole; itraconazole + lactobacilli agent
Drug: lactobacillus gasseri — Lactobacillus vaginal tablets monthly given through 6 days
  Arms: itraconazole + lactobacilli agent
Drug: classic homeopathy (carcinosin M, nux vomica, pulsatilla M, ferrum metallicum, sepia M, etc. as prescribed) — CH treatment was provided by a licensed CH practitioner. Specifically, a personal history was taken and an individualised treatment scheme was prescribed. The most often used homeopathic remedies were carcinosin M, nux vomica, pulsatilla M, ferrum metallicum, and sepia M. Potencies of homeopathic remedies ranged from C 30 to C 1000.
  Arms: classic homeopathy (CH)

SUMMARY:
A prospective study to evaluate the efficacy of classic homeopathic therapy compared to maintenance itraconazole therapy with and without additional exogenous lactobacillus for treatment of recurrent Candida vaginitis.

DETAILED DESCRIPTION:
Objective:

Antimycotics effectively treat sporadic and recurrent vulvovaginal candidiasis (RVVC). Classic homeopathy (CH) is also used to treat this condition. We compared the efficacy of CH and itraconazole in reducing the frequency of RVVC episodes.

Design:

Single-centre, prospective, randomized.

Sample:

One-hundred-and-fifty patients with a history of RVVC and an acute episode of VVC.

Methods:

Women were randomised into 3 groups: itraconazole with lactobacilli (group 1), itraconazole without lactobacilli (group 2) and CH (group 3). Itraconazole treatment of acute infection was followed by a 6-months maintenance regimen with monthly single-day itraconazole (200 mg bid). Thereafter, patients were followed without treatment for 6 months. Women in group 1 were given additional vaginal lactobacilli for six days per month. CH treatment was performed for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years, premenopausal
* Negative pregnancy test
* Signed informed consent
* At least 4 Episodes of Candidiasis within the last year
* Candida detectable by culture
* Negative Hepatitis- and HIV-Serology
* No Allergy to Itraconazole

Exclusion Criteria:

* Under 18 years

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 144 (Actual)
Dates: Start 2000-05; Primary Completion 2006-02 (Actual); Study Completion 2006-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Armin Witt, MD, Principal Investigator — Vienna Medical School
Locations (1):
- Vienna Medical School, Vienna, Austria

RESULTS

PARTICIPANT FLOW:
Groups:
- Itraconazole: itraconazole alone
- Itraconazole + Lactobacillus Gasseri: itraconazole + local lactobacillus gasseri
Period: Overall Study
Arm/Group | Itraconazole | Itraconazole + Lactobacillus Gasseri | Classic Homeopathy
Started | 48 | 50 | 46
Completed | 23 | 25 | 23
Not Completed | 25 | 25 | 23
Not completed — Lost to Follow-up | 25 | 25 | 23

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Itraconazole | Itraconazole + Lactobacillus Gasseri | Classic Homeopathy | Total
Number analyzed (Participants) | 48 | 50 | 46 | 144
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 48 | 50 | 46 | 144
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.5 (7.8) | 30.4 (7.4) | 30.3 (8.0) | 30.4 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 50 | 46 | 144
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Austria | 48 | 50 | 46 | 144

OUTCOME MEASURES:

1. Primary Outcome: Candida Culture Free After Maintenance Therapy
Description: candida culture free (monthly vaginal cultures were obtained)
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | Itraconazole | Itraconazole + Lactobacillus Gasseri | Classic Homeopathy
Number analyzed (Participants) | 23 | 25 | 23
participants | 18 | 19 | 9

ADVERSE EVENTS:
Time Frame: 12 months
Description: Systematik Assessment by using a questionnaire
Arm/Group | Itraconazole | Itraconazole + Lactobacilli Agent | Classic Homeopathy (CH)
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/50 | 0/46
Other Adverse Events (participants affected / at risk) | 0/48 | 0/50 | 0/46

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes